CLINICAL TRIAL: NCT06946732
Title: Acostream Use in Patients With High Risk and Intermediate-risk Acute Pulmonary Embolism (The ARTIST Study)
Brief Title: Acostream Use in Patients With High Risk and Intermediate-risk Acute Pulmonary Embolism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Xiamen Cardiovascular Hospital, Xiamen University (Other); Nantong University Affiliated Hospital (Unknown); Chengdu University of Traditional Chinese Medicine (Other); Shanghai No.1 Hospital (Unknown); First Affiliated Hospital of Fujian Medical University (Other); Jinhua Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The ARTIST study
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Embolism (PE)
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The Acostream aspiration group (Experimental): The pulmonary thrombus removal by Acostream.
  Interventions: Device: Acostream aspiration

INTERVENTIONS:
Device: Acostream aspiration — The pulmonary thrombus removal by Acostream.

SUMMARY:
The registry is to evaluate the safety and feasibility of catheter-directed aspiration for patients with high-risk and intermediate-high-risk pulmonary embolism using Acostream.

DETAILED DESCRIPTION:
The registry is a prospective, multicenter, observational study involving 130 patients across up to seven sites in China. The aim of this study is to evaluate the safety and feasibility of catheter-directed thrombectomy using Acostream in patients with high-risk and intermediate-high-risk pulmonary embolism. The primary endpoint of the study is the efficacy and safety of pulmonary thrombus removal, assessed by reduction of ventricular strain, decrease in vascular obstruction, overall clinical improvement, and the early mortality rate from pulmonary embolism. Secondary endpoints include the total mortality rate of PE and the incidence of complications in the procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18≤Age≤85
* Clinical symptoms and presentation consistent with pulmonary embolism (PE).
* PE symptoms duration ≤ 14 days.
* High risk PE patients with absolute contraindications to systemic thrombolysis or its failure (refractory circulatory collapse) not eligible for surgical embolectomy.
* Intermediate-high risk PE patients with right ventricle dysfunction (right ventricle/ left ventricle >0.9) confirmed by computed tomography pulmonary angiography or transthoracic echocardiography.

Exclusion Criteria:

* Pregnancy.
* Refusal to sign the informed consent form.
* Presence of intracardiac thrombus.
* Presence of chronic left heart failure with an ejection fraction lower than 30% Diagnosed thrombophilia.
* History of severe or chronic pulmonary hypertension.
* Serum creatinine level higher than 1.8 mg/dl.
* Known serious and uncontrolled sensitivity to radiographic agents.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of RV/LV | 48 hours
  The ratio of right ventricular diameter to left ventricular diameter (RV/LV) decreased compared to baseline

SECONDARY OUTCOMES:
Surgical success rate | Immediately after surgery
Changes in pulmonary artery pressure before and after surgery | 48 hours
Changes in arterial oxygen pressure before and after surgery | 14 days
Clinical deterioration incidence | 48 hours
  Clinical deterioration incidence includes tracheal intubation, mechanical ventilation, arterial hypotension>1 hour or shock, cardiopulmonary resuscitation, significant deterioration of oxygenation, and emergency surgical thrombectomy)
All-cause mortality rate | 1, 3, 6, 12 months
Symptomatic PE recurrence rate | 1, 3, 6, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided